CLINICAL TRIAL: NCT03328767
Title: A Pilot Randomised Controlled Trial in Extracorporeal Membrane Oxygenation Physical Training (ECMO-PT)
Brief Title: Extracorporeal Membrane Oxygenation Physical Training
Acronym: ECMO-PT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: Toronto General Hospital (Other); Monash University (Other); The Alfred (Other); Royal Prince Alfred Hospital, Sydney, Australia (Other); The Prince Charles Hospital (Other Government); St Vincent's Hospital, Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANZICRC/ECMO/001
Record Dates: First submitted 2017-10-24; First posted 2017-11-01 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Critically Ill, Mechanically Ventilated; Extracorporeal Membrane Oxygenation Complication
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: A 30 patient, multicentre, randomised, trial of early individualised physical training compared to standard care.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early activity and Mobilisation intervention (Experimental): Patients will be randomised within 48 hrs of commencing ECMO. Patients unable to initially receive active physical training will receive passive physical training for a minimum of 20 minutes and a maximum of one hour per day to maintain joint and muscle activity until active physical training is commenced. The intervention involves a progression of exercises with the objective of rehabilitating the patient at the highest level of exercise possible for the patient for the longest period of time that can be tolerated (up to 60 minutes) at each session, based on our published ICU mobility scale now used internationally in ICU trials. This is performed with or without IMV (including both endotracheal tubes or tracheostomies).
  Interventions: Behavioral: Early activity and Mobilisation intervention
- Standard Care (No Intervention): The control group will receive standard care from physiotherapy staff not involved in delivering the intervention. We have previously established that standard care in Australia for a patient receiving prolonged IMV (control group intervention) frequently involves no active exercise out of bed.

INTERVENTIONS:
Behavioral: Early activity and Mobilisation intervention — The early activity and mobilisation intervention is comprised of exercises based on a reproducible, physiological approach using both strength and functional activities
  Arms: Early activity and Mobilisation intervention

SUMMARY:
Critically ill patients who require extracorporeal membrane oxygenation (ECMO) are the sickest in the hospital. More patients are surviving but survivors have compromised functional recovery for months or years. This trial aims to determine if early, physical training commenced within 48 hours of ECMO is feasible and improves muscle strength and functional status in patients compared to standard practice in a randomised controlled trial of 30 ICU patients.

DETAILED DESCRIPTION:
The use of extracorporeal membrane oxygenation (ECMO) has expanded dramatically in Australia and globally. While life-saving in the short-term, it is typically associated with prolonged immobility and inflammation, which contributes to severe muscle weakness and wasting. Standard care delivers minimal physical training while patients remain on ECMO because standard care prioritises concerns about catheter dislodgement and cardio-respiratory strain. However, in other intensive care unit (ICU) conditions, techniques have been developed to allow early physical training in patients previously thought too unstable to be exercised, with important patient-centred and long-term cost-saving benefits. Our preliminary work shows that early individualised physical training is safe in ICU patients. A multicentre pilot study to establish feasibility in ECMO patients is urgently needed.

The primary aim is to test the hypothesis that early, individualised, physical training (commenced within first 48 hours of ECMO) is feasible and improves functional recovery (the highest level of activity and duration). This has previously been reported to be associated with improved independent function at hospital discharge and discharge to home.1 The secondary aims are to test the hypothesis that early individualised physical training is (i) safe; (ii) improves muscle strength at day 7 and 10 and 20; and (iii) improves functional status (IMS) at day 7, 10 and 20 in ECMO patients relative to standard care.

We are also aiming to describe the acute physiological effects of early physical training (commenced within 48hours of ECMO initiation) Respiratory and haemodynamic parameters, along with ECMO settings, will be recorded 30 minutes prior to each physical training session, during the session and 30 minutes post the training session. In addition, the range of values (min to max) for these parameters will be recorded for each 24hour period over the 7 days.

ELIGIBILITY:
Inclusion Criteria:

* adults ≥ 18 years of age
* were physically independent prior to the current admission;
* receiving ECMO (veno-arterial or veno-venous) for at least 24 hours;
* clinician in charge of patient care has no objection to randomisation

Exclusion Criteria:

* have been in ICU > 5 days prior to the commencement of ECMO;
* have received ECMO for more than 48 hours;
* in the opinion of the treating clinician, is not expected to recover in 90 days (e.g. intracerebral haemorrhage);
* whom death is expected within 24 hours;
* are unable to communicate in English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of delivering the intervention in the first 7 days after randomisation and the separation between the groups | 7 days
  Feasibility of delivering the intervention in the first 7 days after randomisation and the separation between the groups using the ICU mobility scale to report the highest level of activity. It is reported as median (IQR) over 7 days.

SECONDARY OUTCOMES:
Time to first stand out of bed | Within the first 28 days
  Time to first stand out of bed (within the first 28 days)
Incidence of Treatment-Emergent Adverse Events, Safety events (including decannulation of ventilator or ECMO cannula, fall to the floor during mobilization, desaturation SpO2 < 85%) at anytime during the first 7 days | During the first 7 days
  Incidence of Treatment-Emergent Adverse Events, Safety events (including decannulation of ventilator or ECMO cannula, fall to the floor during mobilization, desaturation SpO2 < 85%) at anytime during the first 7 days
Strength at day 7 and 10 | Days 7 & 10
  Strength at day 7 and 10
Function (reported as ICU mobility scale) measured at days 7, 10 and 20 | Days 7, 10 & 20
  Function (reported as ICU mobility scale) measured at days 7, 10 and 20
ICU and hospital length of stay | Time from ICU admission to ICU and hospital discharge respectively censored at day 90
  ICU and hospital length of stay (time from ICU admission to ICU and hospital discharge respectively censored at day 90)
ICU and in-hospital mortality | Time from ICU admission to ICU and hospital discharge respectively censored at day 90
  ICU and in-hospital mortality (time from ICU admission to ICU and hospital discharge respectively censored at day 90)

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (4):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St Vincent's Hospital, Sydney, New South Wales
  - The Prince Charles Hospital, Chermside West, Queensland
  - Alfred Hospital, Melbourne, Victoria
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Yes

REFERENCES:
- [Background] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M. Developing and evaluating complex interventions: the new Medical Research Council guidance. Int J Nurs Stud. 2013 May;50(5):587-92. doi: 10.1016/j.ijnurstu.2012.09.010. Epub 2012 Nov 15. No abstract available. PMID 23159157
- [Background] Hodgson C, Needham D, Haines K, Bailey M, Ward A, Harrold M, Young P, Zanni J, Buhr H, Higgins A, Presneill J, Berney S. Feasibility and inter-rater reliability of the ICU Mobility Scale. Heart Lung. 2014 Jan-Feb;43(1):19-24. doi: 10.1016/j.hrtlng.2013.11.003. Epub 2013 Nov 19. PMID 24373338
- [Background] Tipping CJ, Bailey MJ, Bellomo R, Berney S, Buhr H, Denehy L, Harrold M, Holland A, Higgins AM, Iwashyna TJ, Needham D, Presneill J, Saxena M, Skinner EH, Webb S, Young P, Zanni J, Hodgson CL. The ICU Mobility Scale Has Construct and Predictive Validity and Is Responsive. A Multicenter Observational Study. Ann Am Thorac Soc. 2016 Jun;13(6):887-93. doi: 10.1513/AnnalsATS.201510-717OC. PMID 27015233
- [Background] Borg G. Ratings of perceived exertion and heart rates during short-term cycle exercise and their use in a new cycling strength test. Int J Sports Med. 1982 Aug;3(3):153-8. doi: 10.1055/s-2008-1026080. PMID 7129724
- [Background] Berney S, Haines K, Skinner EH, Denehy L. Safety and feasibility of an exercise prescription approach to rehabilitation across the continuum of care for survivors of critical illness. Phys Ther. 2012 Dec;92(12):1524-35. doi: 10.2522/ptj.20110406. Epub 2012 Aug 9. PMID 22879441
- [Background] Hodgson CL, Stiller K, Needham DM, Tipping CJ, Harrold M, Baldwin CE, Bradley S, Berney S, Caruana LR, Elliott D, Green M, Haines K, Higgins AM, Kaukonen KM, Leditschke IA, Nickels MR, Paratz J, Patman S, Skinner EH, Young PJ, Zanni JM, Denehy L, Webb SA. Expert consensus and recommendations on safety criteria for active mobilization of mechanically ventilated critically ill adults. Crit Care. 2014 Dec 4;18(6):658. doi: 10.1186/s13054-014-0658-y. PMID 25475522
- [Background] Puthucheary ZA, Denehy L. Exercise Interventions in Critical Illness Survivors: Understanding Inclusion and Stratification Criteria. Am J Respir Crit Care Med. 2015 Jun 15;191(12):1464-7. doi: 10.1164/rccm.201410-1907LE. No abstract available. PMID 26075426
- [Derived] ECMO-PT Study Investigators; International ECMO Network. Early mobilisation during extracorporeal membrane oxygenation was safe and feasible: a pilot randomised controlled trial. Intensive Care Med. 2020 May;46(5):1057-1059. doi: 10.1007/s00134-020-05994-8. Epub 2020 Mar 16. No abstract available. PMID 32179935
- See also: Early mobilisation during extracorporeal membrane oxygenation was safe and feasible: a pilot randomised controlled trial — https://doi.org/10.1007/s00134-020-05994-8